CLINICAL TRIAL: NCT01713881
Title: Effect of a Tracking Program on Colon Adenoma Surveillance and Adherence to Guideline Recommendations
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, R. Keith Fincher, MD, FACP, FACG, Gastroenterologist, United States Department of Defense
Other Study IDs: DDEAMC-Fincher 1
Record Dates: First submitted 2012-10-23; First posted 2012-10-25 (Estimated); Last update posted 2014-03-20 (Estimated); Status verified 2014-03

CONDITIONS: Colon Polyp Surveillance
Keywords: Polyp; colonoscopy; surveillance
MeSH Terms: conditions — Polyps

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- post-registry: Registry Group:
  * Select 500 consecutive patients from the polyp registry who were found to have a tubular adenoma on a colonoscopy done between 2007-2008 from the polyp registry.
  * Quantify the completion rate and time between index and surveillance colonoscopy after the establishment of the polyp surveillance program (2006-2013).
- pre-registry: Pre-registry Group: Select 380 consecutive patients who were found to have a tubular adenoma on a colonoscopy done between April 2004-Nov 2006.

SUMMARY:
This will be a retrospective chart review of 880-1000 patients who had a colonoscopy and were found to have a tubular adenoma between the years of 2004-2008. We will compare the rate and timing of completion of repeat colonoscopies pre and post establishment of a polyp registry (tracking system) in 2006. Each group will be composed of up to 500 subjects consecutively identified from all the patients who underwent colonoscopy and were found to have a tubular adenoma (Group 1-2004 to 2006, Group 2 2007-2008).

DETAILED DESCRIPTION:
This will be a retrospective chart review of 880-1000 patients who had a colonoscopy and were found to have a tubular adenoma between the years of 2004-2008. We will compare the rate and timing of completion of repeat colonoscopies pre and post establishment of a polyp registry (tracking system) in 2006. Each group will be composed of 380-500 subjects consecutively identified from all the patients who underwent colonoscopy and were found to have a tubular adenoma (Group 1-2004 to 2006, Group 2 2007-2008).

ELIGIBILITY:
Inclusion Criteria:

* Any adenoma found on screening/surveillance colonoscopy (ICD9-211.3, Procedure code 45385 or 45380)
* Greater than 18 years old

Exclusion Criteria:

* Less than 18 years old
* Diagnosis of IBD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with colon polyps
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2012-08; Primary Completion 2013-12 (Actual); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Percentage completing follow up colonoscopy | 12 months
  A polyp tracking program (registry) decreases the amount of patients lost to follow up.

CONTACTS AND LOCATIONS:
Locations (1):
- D.D. Eisenhower Army Medical Center, Fort Gordon, Georgia, United States